CLINICAL TRIAL: NCT05267496
Title: Effect of Oscillating Positive Expiratory Pressure Therapy on the Frequency of Pulmonary Atelectasis in Thoracic Cancer Patients Undergoing Chest Surgery
Brief Title: Oscillating Positive Expiratory Pressure Therapy for Patients With Thoracic Neoplasms Undergoing Chest Surgery
Acronym: AEROBIKA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Nacional de Cancerologia de Mexico (Other)
Responsible Party: Principal Investigator, Oscar Gerardo Arrieta Rodríguez, Coordinator of the Thoracic Oncology Unit, Instituto Nacional de Cancerologia de Mexico
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CEI/1417/19
Record Dates: First submitted 2022-02-24; First posted 2022-03-04 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Lung Cancer; Mediastinal Tumor; Pleural Tumor
MeSH Terms: conditions — Lung Neoplasms; Mediastinal Neoplasms; Pleural Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional rehabilitation (Other): Patients will receive conventional pulmonary rehabilitation
  Interventions: Procedure: Pulmonary rehabilitation
- AEROBIKA (Experimental): Patients will receive conventional pulmonary rehabilitation in addition to an oscillating positive expiratory pressure device
  Interventions: Device: oscillating positive expiratory pressure device; Procedure: Pulmonary rehabilitation

INTERVENTIONS:
Device: oscillating positive expiratory pressure device — Patients randomized to the experimental arm of the study will receive an AEROBIKA oscillating positive expiratory pressure device in addition to the standard pulmonary rehabilitation program. The patient will receive instructions pertaining to the use of the device during the first evaluation visit to the rehabilitation service and this information will be reinforced at each follow-up visit. The patient will receive a log book in order to record date and time of use to assess treatment compliance and an instructions and maintenance booklet will be handed out to ensure adequate use of the device.
  Other Names: AEROBIKA
  Arms: AEROBIKA
Procedure: Pulmonary rehabilitation — Educational ventilatory techniques will be explained in order to re-educate respiratory muscles and increase patient awareness regarding the importance of complying with the exercise schedule to improve muscular strength. Including:
  Pre-surgical rehabilitation
  * Directed ventilation
  * Physical conditioning Post-surgical rehabilitation
  * Diaphragmatic mobilization
  * Thoracic expansion through incentive flow spirometry

SUMMARY:
This randomized clinical study aims to assess the use of an oscillating positive expiratory pressure device (AEROBIKA) in patients with thoracic neoplasms who undergo chest surgery.

The main questions it aims to answer are:

If the use of the AEROBIKA device reduces the incidence of atelectasis in oncological patients undergoing lung resection.

If the use of the AEROBIKA device reduces hospital readmission and days of hospital stay.

Participants who accept to participate will be sorted to receive a conventional rehab therapy (group A), otherwise a conventional rehab therapy plus AEROBIKA device (group B).

Researchers will compare patients from group A versus group B to see if patients develop atelectasis.

DETAILED DESCRIPTION:
Clinical evaluation

1. At patients´ first visit, demographic, clinical, and imaging variables will be obtained from INCan medical history and electronic record.
2. The patient will be called one week before the date of surgery to the Pulmonary Rehabilitation service. Evaluation of lung function will be carried out through tests by means of spirometry, oscilometry, gas exchange with oxygen saturation measurement and a submaximal exercise test which is the 6 minute walk. Tests will be performed at the following times: before surgery (basal) and after surgery (one month, 2 months and 3 months).
3. The EORTC, QLQ-C30 and QLQ LC13 quality of life questionnaires and a respiratory symptom questionnaire, St. George, will be performed at the same time (before surgery and after surgery (per month, 2 months and 3 months).
4. Patients will be referred to the Lung Rehabilitation Service and a respiratory rehabilitation programme will be initiated. All patients, regardless of the assigned group will carry out a conventional rehabilitation program which consists of TWO PHASES (Pre-surgical Rehabilitation and Post-surgical Rehabilitation).

INTERVENTION GROUP

1. At the first visit to the Pulmonary Rehabilitation service, the patient in the intervention group will receive an AEROBIKA device, at no cost, which the patient can take home.
2. The patient will be instructed on the use of the device by the lung rehabilitation service and knowledge will be reinforced at each visit.
3. The patient will place the date and time of use to assess adherence to treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a confirmed diagnosis of lung cancer, mediastinal tumors or mesothelioma who are candidates for surgical resection through thoracotomy or sternotomy.
2. Measurable disease
3. Age from 18 to 75 years
4. Peak Expiratory flow of 10 liters/min
5. Eastern Cooperative Oncology Group (ECOG) performance status 0-2
6. Karnofsky score 70-100
7. Patients willing and able to comply with all study procedures and follow-up visits.
8. Patients who agree to participate and sign an informed consent form

Exclusion Criteria:

1. Unstable systemic disease, including active infection, cardiac or hemodynamic diseases or neurological diseases.
2. Patients with cognitive impairment who are not able to perform the pulmonary rehabilitation exercises.
3. Oral cavity or facial trauma.
4. Esophagus surgery
5. Active hemoptysis
6. Tympanic rupture or middle ear pathology.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2019-08-13 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Reduction of lung atelectasis | Radiographs will be taken after 3 months of surgery
  The reduction of atelectasis will be assessed according to a visual examination of thoracic radiography.
  In radiography, it is defined as a reduction of lung volume accompanied by an increase in opacity (radiography) or attenuation (CT) in the affected portion of the lung. Atelectasis is often associated with displacement of the cisura, bronchi, vessels, diaphragm, heart, or mediastinum. The distribution can be lobar, segmental, or subsegmental. They are classified: as linear, discoid, or platellary.

CONTACTS AND LOCATIONS:
Overall Officials: Oscar Arrieta, MD,MSc, Principal Investigator — Instituto Nacional de Cancerología de México
Locations (1):
- Instituto Nacional de Cancerologia, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No